CLINICAL TRIAL: NCT04063358
Title: Timing of Anti-vascular Endothelial Growth Factor（Anti-VEGF） Intravitreous Injections for Diabetic Macular Edema(DME) in Patients Undergoing Cataract Surgery
Brief Title: Anti-VEGF Intravitreous Injections for Diabetic Macular Edema in Patients Undergoing Cataract Surgery
Acronym: Anti-VEGF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Military Medical University (Other)
Responsible Party: Principal Investigator, pandongyan, Principal Investigator, Second Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SecondMMU2019
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Diabetic Macular Edema; Cataract
MeSH Terms: conditions — Cataract | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Lucentis injected Pre-operatively (Experimental): Lucentis injected 2 weeks before cataract surgery
  Interventions: Drug: Lucentis
- Lucentis injected intra-operatively (Active Comparator): Lucentis injected during the course of the surgery by cataract surgeon.
  Interventions: Drug: Lucentis
- Lucentis injected post-operatively (Experimental): Lucentis injected 2 weeks after cataract surgery
  Interventions: Drug: Lucentis

INTERVENTIONS:
Drug: Lucentis — Lucentis 0.5 MG Per 0.05 ML Injection

SUMMARY:
The investigators aim to evaluate how different timing of anti-VEGF intravitreous injections affect visual acuity (BCVA) in patients with diabetic macular edema who are undergoing cataract surgery; and to evaluate how different timing of anti-VEGF intravitreous affect OCT CSF thickness and total number of postoperative injections in patients with diabetic macular edema who are undergoing cataract surgery.

DETAILED DESCRIPTION:
Cataract is very common in diabetic patients and can lead to significant vision loss and disability without medical intervention. Diabetic patients, particularly those with diabetic macular edema (DME), experience poorer visual outcomes after undergoing cataract surgery compared to non-diabetics. An increased risk in the development of post-operative cystoid macular edema and exacerbation of baseline DME is reported and this poses a significant challenge in managing concomitant DME and visually-significant cataracts.

Goals of the study are to evaluate how different timing of anti-VEGF intravitreous injections (before operation, intra-operation or after-operation) affect visual acuity (BCVA) in patients with persistent diabetic macular edema who are undergoing cataract surgery; and to evaluate how different timing of anti-VEGF intravitreous injections affect OCT CSF thickness and total number of postoperative injections in patients with diabetic macular edema who are undergoing cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

Adults over age 18 with diabetes mellitus, diabetic macular edema and visually significant cataracts planning to undergo cataract surgery

Exclusion Criteria:

Patients who have undergone panretinal photocoagulation (PRP) in prior 4 months or an ocular condition (other than cataract and DME) that might affect visual acuity during course of study.

Patients with history of vitrectomy. Patients with neovascular glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-08-22 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in best-corrected visual acuity (BCVA) | 1 month, 3 months , 6 months and 12 months after cataract surgery
  BCVA is a measurement of the best vision correction that can be achieved, such as glasses, as measured on the standard Snellen eye chart. For example, if uncorrected eyesight is 20/200, but patient can see 20/20 with glasses, the BCVA is 20/20.
Change in optical coherence tomography (OCT) central subfield (CSF) thickness | 24 hours post-operatively, 1 month, 3 months , 6 months and 12 months after cataract surgery
  Optical coherence tomography (OCT) is an important imaging modality in the evaluation and management of retinal diseases. Change in central subfield (CSF) thickness will be measured and recorded.

SECONDARY OUTCOMES:
Total number of postoperative injections | 12 months after cataract surgery
  Total number of postoperative injections will be calculated
percentage of patients with diabetic retinopathy progression | 12 months after cataract surgery
  patients with diabetic retinopathy progression will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: wei shen, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No